CLINICAL TRIAL: NCT03034369
Title: Caring for the Whole Person: A Patient-Centered Assessment of Integrated Care Models in Vulnerable Populations
Brief Title: Caring for the Whole Person
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Providence Health & Services (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Oregon Health and Science University (Other); Cascadia Addiction Research and Education, LLC (Unknown); Umpqua Community Health Center (Unknown); Mosaic Medical (Unknown); North Portland Clinic (Unknown); Providence Medical Group (Unknown); Rockwood Clinic (Unknown); The Bend Clinic (Unknown); Yamhill CCO (Unknown); The Annex (Unknown); Cascadia Gardiner Clinic (Unknown); Umpqua Expanded Care Clinic (Unknown); Bridges Clinic (Unknown)
Responsible Party: Sponsor
Other Study IDs: 14-247A
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Behavioral Health
Keywords: Integration; Primary Care; Behavioral Health; Health Care Reform; Medical Home; Accountable Care Organization
MeSH Terms: interventions — Health Services Accessibility

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Safety Net Clinic Patients: A Cohort of patients in 12 different primary care clinics will be studied to measure how changes in different integration factors impacts the following patient reported outcomes at baseline and 12 months: Access to Care, Patient-Provider Relationship, Patient-Clinic Interactions, Stigma, Provider Continuity, Symptom Severity, Diagnoses, and Social Support. Health care claims data will be accessed to analyze Depression Screening, Preventive Screening, Inpatient Hospitalization Utilization, Inpatient Readmissions, and Post-Admission follow-up at baseline and 12 months.
  Interventions: Other: Access to Care; Other: Depression Screening; Other: Patient-Provider Relationship; Other: Patient-Clinic Interactions; Other: Stigma; Other: Provider Continuity; Other: Symptom Severity; Other: Diagnoses; Other: Social support; Other: Preventive Screening; Other: Inpatient Hospitalization Utilization; Other: Inpatient Readmissions; Other: Post-Admission follow-up

INTERVENTIONS:
Other: Access to Care — Patient reported outcome survey administered at baseline and 12 months to measure satisfaction with access to care.
Other: Depression Screening — Analysis of health care claims data for depression screenings at baseline and 12 months.
Other: Patient-Provider Relationship — Patient reported outcome survey administered at baseline and 12 months to measure satisfaction with patient-provider relationship.
Other: Patient-Clinic Interactions — Patient reported outcome survey administered at baseline and 12 months to measure satisfaction with patient-clinic interactions.
Other: Stigma — Patient reported outcome survey administered at baseline and 12 months to measure perceived stigma.
Other: Provider Continuity — Patient reported outcome survey administered at baseline and 12 months to measure satisfaction with provider continuity.
Other: Symptom Severity — Patient reported outcome survey administered at baseline and 12 months to measure symptom severity.
Other: Diagnoses — Patient reported outcome survey administered at baseline and 12 months to measure diagnoses.
Other: Social support — Patient reported outcome survey administered at baseline and 12 months to assess social support and outlets.
Other: Preventive Screening — Analysis of health care claims data for preventive screenings at baseline and 12 months.
Other: Inpatient Hospitalization Utilization — Analysis of health care claims data for Inpatient Hospitalization Utilization at baseline and 12 months.
Other: Inpatient Readmissions — Analysis of health care claims data for Inpatient Hospitalization Readmissions at baseline and 12 months.
Other: Post-Admission follow-up — Analysis of health care claims data for Post-Admission follow-up at baseline and 12 months.

SUMMARY:
The goal of this study is to identify outcomes associated with Behavioral Health Integration (BHI) that matter to patients, to compare changes in outcome over time to measure the impact of different BHI models on different patients, and to create and maintain an Integration Learning Collaborative.

DETAILED DESCRIPTION:
Twelve safety net clinics have been selected to be a part of this study. The clinics vary on a BHI continuum level, which includes minimal collaboration, basic collaboration at a distance, basic collaboration on site, close collaboration (partially integrated) and close collaboration (fully integrated).

Twelve-thousand patients will be randomly selected from the 12 clinics to be invited to participate in the study. Patients who elect to participate will complete a survey at baseline to collect patient-reported outcomes and again twelve months later.

The Oregon All Providers All Claims (APAC) database will be accessed to analyze financial data regarding the patients at baseline and 12 months.

The hypothesis is that the degree of clinic BHI will predict patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18
* Received care at a safety net care clinic in Oregon

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients accessing care at safety net clinic in Oregon.
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in patient reported outcomes | 12 months
  Change in patient reported outcomes at baseline and 12 months
Change in health care claims | 12 months
  change in health care claims at baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bill J. Wright, PhD, Principal Investigator — Director, Center for Outcomes Evaluate and Education, Providence Health & Services
Locations (1):
- Center for Outcomes Research and Education, Providence Health & Services, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Center for Outcomes Research and Education, Providence Health & Services — http://oregon.providence.org/our-services/c/center-for-outcomes-research-and-education-core/